CLINICAL TRIAL: NCT04935255
Title: Determining the Clinical Relevance of the inTeraction Between AprepitaNt aNd EtoposiDe; an Observational Pharmacokinetic Study
Brief Title: Determining the Clinical Relevance of the inTeraction Between AprepitaNt aNd EtoposiDe
Acronym: TANNED
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TANNED
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Testicular Cancer
Keywords: aprepitant; etoposide; pharmacokinetic interaction; CYP3A4; clinical relevant interaction; pharmacokinetics
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: The participating patients are treated according to local standard treatment (consisting of etoposide 100mg/m2 and cisplatin 20 mg/m2 during 5 consecutive days). Anti-emetic treatment with aprepitant will be given during days 3 to 7.
  Interventions: Other: Blood sampling - Pharmacokinetic assessment

INTERVENTIONS:
Other: Blood sampling - Pharmacokinetic assessment — Two pharmacokinetic assessments will be performed (on day 2 and day 4). Each pharmacokinetic assessment consists of 10 samples (5 ml blood).

SUMMARY:
Rationale: In pharmacokinetic studies, aprepitant was shown to be a moderate inhibitor of CYP3A4 activity. Etoposide is metabolised by CYP3A4.

Objective: to investigate the absence of a clinical relevant interaction between aprepitant and etoposide in TC patients treated with (B)EP.

Study design: A single centre, prospective, paired observational pharmacokinetic study in 12 patients with TC who are treated with etoposide during 5 days in combination with cisplatin with or without bleomycin conform the standard BEP or EP-protocol and who will be treated with aprepitant from day 3 until day 7 according to the routine antiemetic protocol. The effect of aprepitant on etoposide will be investigated within the same patient. In this study the patient will serve as its own control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TC who will start or already started treatment with (B)EP
* Age of at least 18 years
* Patients from whom it is possible to collect blood samples
* Patients who are able and willing to give written informed consent prior to screening

Exclusion Criteria:

* Patients who are co-treated with drugs that could interfere with the metabolism of etoposide (including drugs classified as a weak, moderate or strong CYP3A4 inhibitor OR weak, moderate and strong inducers of CYP3A4 according to the table based on the Flockhart table (Appendix 1) less than 30 days prior to study or during the study.
* Creatininclearance <40 ml/min
* Severe liver dysfunction (bilirubin>ULN)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will exist of patients treated at the Radboudumc who are diagnosed with TC and are treated with (B)EP according to standard treatment guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Exposure to etoposide | 24 hours after administration
  Etoposide exposure (AUC0-24hr) with and without cotreatment with aprepitant

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud UMC, Nijmegen, Netherlands